CLINICAL TRIAL: NCT00705952
Title: Effect of Intensive Lifestyle Intervention on Hormonal Factors Regulating Food Intake and Blood Glucose Control in Patients With New Onset Type 2 Diabetes.
Brief Title: Group Lifestyle Intervention for People With New Onset Type 2 Diabetes.
Acronym: GLP4Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Professor David Kerr, Royal Bournemouth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP4Health ("GLP-1"); REC ref.: 07/H0201/100
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes
Keywords: No diabetes medications; New onset
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — Diet, exercise and behavioural change intervention.

SUMMARY:
The purpose of the study is to assess whether weight loss achieved through a programme of intensive lifestyle management can result in enhanced production of Glucagon-Like Peptide-1 (GLP-1) together with improvements in the release of insulin and glucagon and thus improvements in glycaemic control (HbA1c), in patients with new onset type 2 diabetes.

This is a cohort study with comparisons made between assessments at baseline, after an initial four months of intensive intervention and after a further four months follow up (maintenance period). Each patient will participate in the study for 8 month. The entire study period will be 24 months.

All patients with new onset type 2 diabetes (within 2 weeks of diagnosis) will be recruited from those referred to the Type 2 Diabetes Education Programme in the community ("FOCUS"), as per standard practice. The investigators will also hope to recruit direct from local GP surgeries who will be advised of the study. At this point, patients will be given a study information sheet with a contact number if they wish to participate in the study.

Individuals who are unable to give consent, who would be unable to attend all the programme sessions for medical or other reasons, who are prescribed oral hypoglycaemic, antiobesity or any other prescription medications that may interfere with the study results or whose BMI is < 25, will be excluded. The investigators will also exclude those who cannot converse competently in English as special arrangements would need to be made for such people attending the programme and this would be impractical in a group setting.

Those willing to participate will be invited for an individual appointment with the dietitian, during which the study structure, aims and procedures will be explained and consent to participate in the study will be obtained. For the first session of the programme, participants will be asked to attend following an overnight fast. Blood samples will be taken for basal measurement of glucose, HbA1c, lipids, insulin, glucagon, GLP-1, leptin, ghrelin and adiponectin. They will then be given a standard 75 g glucose load and sampling repeated at 30 mins (for peak GLP-1 levels). Baseline measurements of weight, height, percent body fat, waistline circumference and blood pressure will also be taken during this session. Following the assessment, patients will participate in the first session of the education programme. The full assessment will be repeated at 4 and 8 months intervals.

The weight management programme will be run by the Specialist Dietitian. It will consist of 2 phases: an initial 4 month intensive weight loss phase, followed by a 4 month weight loss / maintenance phase. The initial four month programme will consist of 8 group education sessions and at least 3 phone calls. The following 4 month programme will consist of 5 group sessions, at least 3 phone calls and 1 individual appointment. Each education session will last 60min. Before the 1st session and, at 4 month and 8 month sessions, bloods will be taken, as above. Before the rest of the sessions, there will be 15 minutes devoted to weight assessment. The programme will be based on portion control and healthy eating and will be supported by behavioural and cognitive change interventions. Such interventions will include self monitoring, stimulus control, goal setting, problem solving and relapse prevention. The specialists from "Bournemouth HealthLink" (a partnership backed by the local NHS, Council and University) will take part in helping participants to increase their activity levels.

The aim is to achieve weight loss of 5% over the first 4 months with, as a minimum, weight maintenance or possible further reduction over the subsequent four months.

DETAILED DESCRIPTION:
The early management of type 2 diabetes usually consists of education related to lifestyle changes especially as 80 to 90% of people with type 2 diabetes are obese. Obesity worsens the metabolic and physiological abnormalities associated with diabetes particularly hyperglycaemia (raised blood sugar), hyperlipidaemia (raised fats in the blood), and hypertension which are prerequisites for macrovascular complications. On the other hand, weight loss is one of the cornerstones of diabetes management as it improves glycaemic (blood glucose) control, lowers triglycerides (a fat in the blood) and low-density lipoprotein cholesterol (the "bad" form of cholesterol) levels and improves blood pressure, mental health and quality of life.

In 1993 the investigators established a structured education programme for patients with new onset type 2 diabetes; following the diagnosis being made in primary care individuals are seen within one week at a nurse led, open-access programme. Since 1994, there has been a 2.5 fold increase in the number of patients diagnosed with type 2 diabetes in our area. At diagnosis, Body Mass Index (BMI) has risen from 28.5 to 31.1kg/m2 associated with a fall in HbA1c (a blood test which gives a measure of long term control of diabetes) levels from 10.3% to 8.1% at presentation. The lower HbA1c at diagnosis probably reflects earlier detection and awareness of the condition. Since 2006, responsibility for providing the education has been transferred to primary care.

More recently, a secondary care based dietitian led group weight management programme comprising more intensive education sessions and regular phone contact was piloted in this unit. A recent evaluation of this service of fifty one overweight and obese individuals who completed the 3-month programme. Average weight loss at 3 months was 4.8 kg equivalent to 4.5 % baseline body weight. Follow up at six months, without further intervention, showed that this was maintained (weight loss 5.8 kg, equivalent to 5.3 %, ns compared to 3/12). 43% of participants achieved >5% weight reduction with 6% achieving >10%. The intervention resulted in significant reduction in waistline circumferences, body fat mass, total cholesterol, HbA1c, fasting blood glucose, and blood pressure.

A number of neuro-endocrine factors (hormones that influences the activity of the brain or nervous system) have a role in the control of insulin secretion and in the regulation of food intake. Glucagon-like peptide-1 (GLP-1) is an incretin hormone, the name based on the observation that the insulin response to an oral glucose load was greater than that following the intravenous administration of an equivalent amount of glucose. Incretin hormones are secreted from the small intestine in response to the presence of nutrients in the intestinal lumen. Physiologically, GLP-1 enhances glucose-mediated insulin secretion and suppresses glucagon (a hormone that opposes the action of insulin) secretion. GLP-1 also induces satiety and improves gastric emptying. In studies of patients with established diabetes, GLP-1 levels and the response to oral glucose have been shown to be attenuated and administration of GLP-1 has normalized both fasting and post-prandial glucose levels. It remains uncertain whether lower GLP-1 levels in established diabetes contribute to the pathogenesis of the condition or are a consequence of chronic hyperglycaemia, though the observation that GLP-1 levels are lower in obese subjects suggests the possibility that the former may be the case.

Recently, the investigators measured GLP-1 levels in patients with newly diagnosed type 2 diabetes to assess the effect of an initial period of lifestyle and dietary adjustment. In this pilot project 9 newly diagnosed patients (time from diagnosis 25 + 5 days, 4 female with mean BMI 27.6 kg/m2 were compared with 9 age, gender and body weight matched controls. All participants had a 75g oral glucose tolerance test with measurements of glucose, insulin, GLP-1 and glucagon with the diabetic patients having a repeat OGTT after 3 months. Compared with controls, diabetic patients had higher glucagon levels, lower active GLP-1 at baseline before the glucose load although AUC levels were not significantly different. After 3 months lifestyle adjustment, 5 patients had achieved weight loss (0.2 to 5 kg) but 4 had gained weight (2.7 to 6.5 kg), giving an average weight change for the group of 0.8 Kg. A small change in HbA1c was observed (7.31% vs 6.96%, p=0.25). The levels of active GLP-1 were augmented in the diabetic group accompanied by an increase in the insulin response at 30 mins. though glucagon levels were unaltered.

It is unclear whether more intensive lifestyle changes would result in greater improvements in GLP-1 production and thus greater improvements in diabetic control. If GLP-1 production can be enhanced early following diagnosis of diabetes, this may have favorable consequences for the patient, as GLP-1 has been shown in animal studies and in vitro, to have a role in the regulation of beta glucose sensing and proliferation of beta-cells.

A number of other neuroendocrine peptides have regulatory roles in energy homeostasis and may influence insulin secretion and glycaemic control. Leptin is a protein hormone produced by adipose (fat) tissue which has a key role in regulating energy intake and expenditure, a suppressive effect on appetite and an increase in metabolism. Circulating leptin levels reflect body fat mass. Leptin can enter the the Central Nervous System (CNS) at and interact with centres in the regulation of appetite and metabolism. Despite these suppressive effects, elevated levels have often been noted in obesity, possibly suggesting resistance to the hormone, though may be a result of stimulation by increased insulin levels, which would be expected in obesity. Leptin in turn can inhibit insulin release so a fall in leptin resulting from weight loss may enhance insulin production and may therefore be beneficial in patients with diabetes.

Unlike leptin, ghrelin is an orixigenic (stimulates appetite) hormone which acts via the Growth Hormone secretagogue receptor. It is the only hormone known to stimulate increased feeding and weight gain. Basal plasma levels are increased in malnutrition and decreased in obesity. In some, but not all studies, insulin has been shown to be an inhibitor of ghrelin release. An anticipated rise in ghrelin with weight reduction might offset the effects of lifestyle intervention through stimulation of appetite and increased intake.

Adiponectin is an adipocyte (fat cell) hormone that modulates a number of metabolic processes, including glucose regulation and fatty acid catabolism, and may have a role in the metabolic derangements of type 2 diabetes. Though produced in adipose (fat) tissue, plasma adiponectin levels are decreased in obesity as a consequence of down regulation. Adiponectin has insulin sensitizing effects and has central effects on energy homeostasis, promoting weight reduction. Levels of adiponectin have been found to be reduced in type 2 diabetes compared with non-diabetic controls. Weight reduction can increase circulating levels. Again little is known about the effect of changes in adiponectin in the early stages of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. New onset of Type 2 Diabetes.
2. BMI>25kg/m2

Exclusion Criteria:

1. Antiobesity, oral hypoglycaemic medications or any other prescription medications that may interfere with the study results
2. Pregnancy
3. Unable to converse competently in English as special arrangements would need to be made for such people and this would be impractical in a group setting
4. Attending another weight management programme
5. Patients who would be unable to attend all the programme sessions for medical or other reasons
6. Any patients from groups listed in A24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Whether weight loss achieved through a programme of intensive lifestyle management can result in enhanced production of Glucagon-Like Peptide-1 together with improvements in glycaemic control, in patients with new onset type 2 diabetes. | 8 months lifestyle programme

SECONDARY OUTCOMES:
To examine the changes in hormonal regulators of energy homeostasis (leptin, adiponectin, ghrelin) and cardiovascular risk factors occurring with this intervention. | 8 months lifestyle programme

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, professor, Principal Investigator — Royal Bournemouth Hospital